CLINICAL TRIAL: NCT04312256
Title: Comparison of Flexor Hallicus Brevis and Adductor Pollicis as Sites for Neuromuscular Monitoring With Electromyography (Thumb vs Great Toe) After Sugammadex Administration
Brief Title: Thumb vs Great Toe Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-011705
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Neuromuscular Blockade; Tetragraph; AMG; EMG
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dominant Hand and great toe (Experimental): Subject scheduled to undergo an elective surgical procedure will have TetraGraph device lead placement on the dominant hand and great toe.
  Interventions: Device: TetraGraph

INTERVENTIONS:
Device: TetraGraph — FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin (ECG) electrodes.

SUMMARY:
Researches are comparing the accuracy of measuring muscle relaxation in the thumb versus the great toe.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients undergoing an elective surgical procedure that requires use of non-depolarizing NMBA agents administered intraoperatively.
* Patients with planned administration of sugammadex as a neuromuscular blocking reversal agent.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm or leg into the sterile field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dominant Hand and Great Toe: Subjects who underwent an elective surgical procedure had TetraGraph device lead placement on the dominant hand and great toe.
  TetraGraph: FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin (ECG) electrodes.
Period: Overall Study
Arm/Group | Dominant Hand and Great Toe
Started | 81
Completed | 81
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dominant Hand and Great Toe
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 73
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 81

OUTCOME MEASURES:

1. Primary Outcome: Onset Time of Muscle Relaxation for Flexor Hallucis Brevis (Great Toe) and Adductor Pollicis (Thumb) Muscles
Description: The amount of time before initial muscle relaxation is recorded via neurostimulation with the Tetragraph device. As measure in seconds.
Time Frame: Up to 1 hour postoperatively
Measure: Median (Full Range); unit: seconds
Groups:
- Flexor Hallucis Brevis (Great Toe): TetraGraph monitoring flexor hallucis brevis (great toe) muscle for all subjects.
- Adductor Pollicis (Thumb): TetraGraph monitoring adductor pollicis (thumb) muscle for all subjects.
Arm/Group | Flexor Hallucis Brevis (Great Toe) | Adductor Pollicis (Thumb)
Number analyzed (Participants) | 81 | 81
seconds | 180.0 [0.0 to 540.0] | 180.0 [0.0 to 840.0]

2. Primary Outcome: Recover Time for Flexor Hallucis Brevis (Great Toe) and Adductor Pollicis (Thumb) Muscles
Description: The amount of time after muscle neurostimulation with the Tetragraph device completion to muscle full recovery. As measure in seconds.
Time Frame: Up to 1 hour postoperatively
Population: Data was not collected nor analyzed in18 subjects great toes. Data was not collected nor analyzed in 13 subjects thumbs.
Measure: Median (Full Range); unit: seconds
Arm/Group | Flexor Hallucis Brevis (Great Toe) | Adductor Pollicis (Thumb)
Number analyzed (Participants) | 63 | 68
seconds | 180 [0.0 to 1020] | 180 [0.0 to 660]

3. Secondary Outcome: Onset Time of Reversal Agent Administered for Flexor Hallucis Brevis (Great Toe) and Adductor Pollicis (Thumb) Muscles
Description: The amount of time from reversal agent administered to initial muscle relaxation increase recorded via neurostimulation with the Tetragraph device. As measure in seconds.
Time Frame: Up to 1 hour postoperatively
Measure: Median (Full Range); unit: seconds
Arm/Group | Flexor Hallucis Brevis (Great Toe) | Adductor Pollicis (Thumb)
Number analyzed (Participants) | 81 | 81
seconds | 180.0 [0.0 to 540.0] | 180.0 [0.0 to 840.0]

4. Secondary Outcome: Recover Time of Reversal Agent Administered for Flexor Hallucis Brevis (Great Toe) and Adductor Pollicis (Thumb) Muscles
Description: The amount of time after reversal agent administered to muscle full recovery recorded via neurostimulation with the Tetragraph device. As measure in seconds.
Time Frame: Up to 1 hour postoperatively
Population: Data was not collected nor analyzed in 18 subjects great toes. Data was not collected nor analyzed in 13 subjects thumbs.
Measure: Median (Full Range); unit: seconds
Arm/Group | Flexor Hallucis Brevis (Great Toe) | Adductor Pollicis (Thumb)
Number analyzed (Participants) | 63 | 68
seconds | 180.0 [0.0 to 1020.0] | 180.0 [0.0 to 660.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately one hour
Arm/Group | Dominant Hand and Great Toe
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04312256/Prot_SAP_000.pdf